CLINICAL TRIAL: NCT06538246
Title: Self-directed Mobile Adaptive Coping Skills Intervention to Improve Psychological Distress Symptoms Among Cardiorespiratory Failure Survivors: Blueprint 2
Brief Title: Adaptive Coping Skills Training to Improve Psychological Distress Among Cardiorespiratory Failure Survivors
Acronym: Blueprint 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Oregon Health and Science University (Other); University of Colorado, Denver (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro00115623
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Depression; Anxiety; Post-traumatic Stress Disorder; Stress; Worries; Pain or Disability; Breath Shortness
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Pain; Dyspnea | interventions — Blueprint Asept; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators will be blinded to group assignment and survey results. Survey results will be reported by the participants via their mobile apps, and so will not be visible to anyone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueprint adaptive coping skills intervention (Experimental): This is a unique adaptive coping skills intervention developed over years of research that targets patients hospitalized for cardiorespiratory conditions. Participants will receive 4 weeks of different Blueprint content through a mobile app. Each week's session includes a within-app HADS survey for safety monitoring. A printed or PDF workbook with complementary content and QR links to app videos is provided.
  Interventions: Behavioral: Blueprint
- Education program control (Active Comparator): This is cardiorespiratory condition-specific content through an iterative process, informed by research on informational needs and past successful education programs. Participants will receive 4 weeks of different 10-minute informational videos unrelated to Blueprint content through a mobile app. Each week's session includes a within-app HADS survey for safety monitoring. A printed or PDF workbook with complementary content and QR links to app videos is provided.
  Interventions: Behavioral: Education program

INTERVENTIONS:
Behavioral: Blueprint — This is a mobile app-based adaptive coping skills intervention that lasts 1 month
  Arms: Blueprint adaptive coping skills intervention
Behavioral: Education program — This is a mobile app-based education program that lasts 1 month
  Arms: Education program control

SUMMARY:
Conditions treated in intensive care units (ICUs) such as the acute respiratory distress syndrome (ARDS), congestive heart failure, COVID pneumonia, and sepsis are common. These can lead to high rates of depression, anxiety, and PTSD that worsen quality of life. Yet there are few effective strategies able to overcome barriers of limited access to mental health care. Even less is known about the experiences of patients from racially and ethnically minoritized populations because of they haven't been included well in past research.

To address this problem, the investigators developed Blueprint, a mobile app that coaches people to use adaptive coping skills to self-manage their symptoms. The investigators found that it reduced depression symptoms and improved quality of life compared to placebo.

To confirm these promising findings, the investigators are doing a formal test of Blueprint. The investigators will enroll 400 people who received ICU care from 4 hospitals (Duke, UCLA, Colorado, and Oregon). These patients will be randomized to receive either the Blueprint mobile app or a special Education Program mobile app the investigators developed. -both delivered through similar mobile app platforms. Our specific aims are to see which program improves symptoms better across 6 months of follow up.

This project addresses national research priorities and could advance the field with a personalizable yet population-focused therapy that could be scaled broadly and efficiently to enhance mental health equity.

DETAILED DESCRIPTION:
Cardiorespiratory conditions such as the acute respiratory distress syndrome (ARDS), congestive heart failure, COVID pneumonia, and sepsis are among the most common causes of mortality and morbidity. They are also notable for high rates of persistent psychological distress symptoms including depression, anxiety, and PTSD that worsen quality of life and outcomes of the underlying conditions. Yet there are few effective strategies able to overcome barriers of limited access to mental health care. Even less is known about distress management among people from structurally disadvantaged backgrounds such as racially and ethnically minoritized populations because of their suboptimal representation in relevant clinical trials.

To fill this gap, the investigators developed Blueprint, an adaptive coping skills training intervention, and have optimized it over years of research. The investigators conducted a multicenter RCT (PCORI PFA 195) of a telephone- and web-based version among those recently hospitalized with serious cardiorespiratory conditions, finding that it reduced depression symptoms and improved quality of life among those with elevated baseline distress. Informed by lessons learned about intervention delivery and eligibility criteria, the investigators next conducted a single-center pilot RCT (R34 HL145387) that targeted a broader population and tested a completely automated, self-guided, symptom-responsive mobile app version of Blueprint. The investigators found excellent adherence and a strong effect on depression, anxiety, PTSD, and quality of life compared to control.

Given these promising findings, a formal test of the Blueprint adaptive coping skills training intervention's efficacy is needed. Therefore, the investigators propose a 5-year multicenter RCT with 6-month follow up in which 400 cardiorespiratory failure survivors with elevated symptoms of psychological distress post-discharge are randomized to either Blueprint or an Education Program control-both delivered through similar mobile app platforms. Our specific aims will: (1) Test Blueprint vs. control on symptoms of depression, anxiety, PTSD, and quality of life; (2) Determine patient-level characteristics associated with a great treatment response among sociodemographic subgroups of interest, also applying a heterogeneity of treatment effects analysis to identify other groups of clinical relevance; and (3) Ensure off-the-shelf intervention readiness for implementation by using an exploratory mixed-methods hybrid type 1 implementation framework analysis that integrates semi-structured interviews with trial participants and quantitative trial data from Aims 1 and 2.

Innovative elements include a fully automated mobile health delivery system that personalizes content in response to changes in symptom trajectories, a focus on racially and ethnically minoritized persons, the integration of a Spanish language intervention version, and strong community engagement. This project addresses national research priorities and could advance the field with a personalizable yet population-focused therapy that could be scaled broadly and efficiently to enhance mental health equity.

ELIGIBILITY:
Inclusion Criteria Inclusion criteria present in the hospital

1. Adult (age ≥18)
2. Managed in an ICU or stepdown unit for ≥24 hours during the time inclusion criterion #3 is met
3. Serious acute cardiorespiratory condition, defined as ≥1 of the following:

   * mechanical ventilation via endotracheal tube for ≥4 hours
   * non-invasive ventilation (CPAP, BiPAP) for ≥4 hours in a 24-hour period provided for acute respiratory failure
   * new use of supplemental oxygen ≥6 liters per minute (or increase in baseline continuous oxygen)
   * use of vasopressors for shock of any etiology
   * use of inotropes for shock of any etiology
   * use of pulmonary vasodilators
   * use of aortic balloon pump or cardiac assist device for cardiogenic shock
   * use of diuretic intravenous drip
   * evidence of acute coronary ischemia (i.e., elevated troponin level, supporting EKG changes, unstable angina symptoms documented)
   * urgent cardiac catheterization
4. Cognitive status intact

   • No history of pre-existing significant cognitive impairment (e.g., dementia) as per medical chart
5. Absence of severe mental illness

   * Treatment for severe mental illness (e.g., psychosis, bipolar affective disorder, schizoaffective disorder, schizoid personality disorder, schizophrenia [as per medical record], hospitalization for any psychiatric disorder) within the 6 months preceding the current hospital admission
   * Evidence of poorly managed severe mental illness
   * No endorsement of suicidality at time of admission or informed consent
6. Functional fluency in English or Spanish (i.e., sufficient knowledge of English or Spanish to complete study tasks like watch videos, complete surveys)

Inclusion criteria present after hospital discharge (i.e., at the time of arrival home after discharge from the hospital)

1. Elevated baseline psychological distress symptoms, defined as a Hospital Anxiety and Distress Scale (HADS) total score ≥8

Exclusion Criteria Exclusion criteria present in the hospital

1. Active alcohol or drug abuse (e.g., admission for alcohol withdrawal, drug-related complication, positive toxicology screening at admission, endorsement of active addiction)
2. Anticipated complex medical needs after discharge that would be disruptive to intervention and follow up; for example:

   * Anticipated surgical procedures
   * Anticipated complex medical regiment (e.g., new chemotherapy, new dialysis, need for repeat surgery, pregnant and near term)
   * Plan for comfort care
3. Other complex needs anticipated that could interfere with the ability to complete study procedures. Examples include:

   * Anticipated disruptive travel
   * Inability to use mobile app
   * Anticipated unstable living situation
4. Anticipated or actual discharge to a location other than independent in a home setting (e.g., nursing home, long-term acute care facility, inpatient rehabilitation facility, home hospice)
5. Persistently impaired cognition as a result of illness (Impairment defined as ≥3 errors on the Callahan cognitive status screen and/or the lack of decisional capacity (i.e., patient could be consented by medical team for a procedure if necessary)
6. Currently imprisoned or incarcerated or in home detention
7. Lack a reliable smartphone with cellular data plan or access to the internet
8. Currently enrolled in another study involving an intervention whose objectives conflict with the objectives of this study
9. Previously enrolled in the trial

Exclusion criteria present after hospital discharge (i.e., at T1 Data Collection conducted at the time of arrival home from the hospital)

1. Failure to randomize within 14 days from planned start date (planned start date is within 3 days post-discharge from the hospital to home to accommodate weekends)
2. Readmission to hospital before randomization completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline, 1 month, 3 months, and 6 months post-randomization
  The HADS evaluates anxiety (7 items) and depression (7 items) with a 14-item instrument assessing symptoms on a 4-point scale rated from 0 "not at all" to 3 "very often indeed". It has a score range of 0 to 42 with higher scores indicating more symptoms.

SECONDARY OUTCOMES:
Post-Traumatic Stress Syndrome inventory (PTSS) | Baseline, 1 month, 3 months, and 6 months post-randomization
  The PTSS rates 10 post-traumatic stress symptoms and has a score range of 10 (no symptoms) to 70 (high burden of symptoms).
EuroQOL-5D visual analog scale (EQ VAS) quality of life measure | Baseline, 1 month, 3 months, and 6 months post-randomization
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' (100) and 'Worst imaginable health state' (0). The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Perceived Stress Scale 4-Item survey (PSS-4) | Baseline, 1 month, 3 months, and 6 months post-randomization
  This is a 4-item short version of the PSS. Scores can range from 0 (lowest stress) to 16 (highest level of stress)

OTHER OUTCOMES:
Patient Health Questionnaire 10-Item symptoms scale (PHQ-10) | Baseline, 1 month, 3 months, and 6 months post-randomization
  The PHQ-10 is an adapted version of the PHQ-15, a measure of physical symptoms. Scores can range from 0 (best) to 30 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cox, Principal Investigator — Professor of Medicine
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share deidentified data via an approved and secure data sharing source on completion of the study and publication of results, as per NIH guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Per NIH guidelines
Access Criteria: To be determined

REFERENCES:
- [Result] Cox CE, Gallis JA, Olsen MK, Porter LS, Gremore T, Greeson JM, Morris C, Moss M, Hough CL. Mobile Mindfulness Intervention for Psychological Distress Among Intensive Care Unit Survivors: A Randomized Clinical Trial. JAMA Intern Med. 2024 Jul 1;184(7):749-759. doi: 10.1001/jamainternmed.2024.0823. PMID 38805199
- [Result] Cox CE, Hough CL, Jones DM, Ungar A, Reagan W, Key MD, Gremore T, Olsen MK, Sanders L, Greeson JM, Porter LS. Effects of mindfulness training programmes delivered by a self-directed mobile app and by telephone compared with an education programme for survivors of critical illness: a pilot randomised clinical trial. Thorax. 2019 Jan;74(1):33-42. doi: 10.1136/thoraxjnl-2017-211264. Epub 2018 May 23. PMID 29793970